CLINICAL TRIAL: NCT07075107
Title: Transcriptomic Analysis (RNAseq) of Blood and Fibroblasts to Establish a Diagnosis in Patients With Rare Diseases
Brief Title: Transcriptomic Analysis of Fibroblasts and Blood in Patients With Rare Diseases
Acronym: ARNseqFibroSan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM23_0469; ID-RCB (Registry Identifier: 2024-A00345-42)
Record Dates: First submitted 2025-05-22; First posted 2025-07-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Rare Genetic Disease
Keywords: genetic analysis by high-throughput DNA sequencing; ARNseq; transcriptomic data; interpretation of sequence variants; Genomic Testing; RNA sequencing data; transcriptome analysis in rare disease; Rare diseases; Intellectual disability
MeSH Terms: conditions — Rare Diseases; Intellectual Disability | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARNseq (Experimental): Patients enrolled in the experimental arm will be seen in consultation to sign the consent form and take samples at one of the participating investigational sites.
  Only one visit is planned as part of the study. This is the inclusion visit, during which skin and blood samples are taken.
  If a pathogenic variant explaining the phenotype is identified in a patient, the clinician following the patient will request confirmation of the variant by targeted analysis (Sanger sequencing) as part of the diagnosis. This result will be returned by the clinician who follows the patient as part of his or her usual care.
  Interventions: Procedure: Blood collection; Procedure: skin biopsy

INTERVENTIONS:
Procedure: Blood collection — Blood is collected in order to perform transcriptomic sequencing from blood
Procedure: skin biopsy — A biopsy of skin is performed in order to perform transcriptomic sequencing on fibroblasts obtained from the biopsy

SUMMARY:
This study aims to answer a key question in the field of rare genetic diseases by determining the prevalence of deleterious variants at RNA level in undiagnosed patients with intellectual disability and/or neonatal hypotonia. This study will put an end to diagnostic erraticism in a number of patients.

Finally, the results of this study will make it possible to compare the two types of tissue used for RNAseq, with a view to facilitating the implementation of this analysis method in the diagnostic setting.

DETAILED DESCRIPTION:
Rationale:

The majority of patients with intellectual disability or neonatal hypotonia remain undiagnosed, despite extensive genetic testing. In fact, standard analyses aimed at detecting abnormalities in the patient's DNA only enable a diagnosis to be made in a third of cases. Our hypothesis is that a certain number of these misdiagnosed patients carry anomalies (pathogenic variants) disrupting the RNA (transcript), which were not identified by DNA sequencing.

This study aims to answer a key question in the field of rare genetic diseases by determining the prevalence of deleterious variants at RNA level in undiagnosed patients with intellectual disability and/or neonatal hypotonia. This study will put an end to diagnostic erraticism in a number of patients.

Finally, the results of this study will make it possible to compare the two types of tissue used for RNAseq, with a view to facilitating the implementation of this analysis method in the diagnostic setting.

Objectives:

Determine the prevalence of variants with a deleterious effect at RNA level, identified by transcriptomic analysis (RNAseq) in diagnostically errant patients with neonatal hypotonia and/or intellectual disability. This analysis will be carried out in parallel on blood and fibroblast culture (skin biopsy).

Compare the number of pathogenic variants identified by RNAseq on blood tissue with the number of pathogenic variants identified by RNAseq on fibroblast culture. The result will help to decide whether a single sample is sufficient to obtain a diagnosis in patients in diagnostic limbo.

Study endpoints:

The number of patients initially in diagnostic errancy in whom a deleterious variant at RNA level was identified by transcriptomic analysis (RNAseq).

The number of deleterious RNA variants identified in patients in diagnostic errancy using ARNseq on fibroblasts and the deleterious RNA variants identified using ARNseq on blood samples.

Study design:

Multicentric descriptive prevalence study

Study Procedures:

Patients (or their parents in the case of minors) will be informed of the possibility of participating in the study during a follow-up consultation as part of their usual care. Patients will also be given a leaflet explaining the study. After a period of reflection, patients will be seen at one of three centers (Marseille, Toulon, Nice) to sign a consent form and take samples.

Only one visit is planned as part of the study. This is the inclusion visit, during which skin and blood samples are taken.

If a pathogenic variant explaining the phenotype is identified in a patient, the patient's physician will request confirmation of the variant by targeted analysis (Sanger sequencing) by the laboratory (Laboratoire de Génétique Moléculaire, APHM) as part of the diagnosis. This result will be provided by the patient's doctor as part of the patient's usual care.

Subjects number: 62

Study Timelines:

Inclusion period: 36 months Duration of follow-up: There is no follow-up for the patient in this study - a single inclusion visit is planned. Results will be reported as part of the patient's usual care.

Duration of analyses: 6 months Total duration (duration of inclusion and duration of analysis): 42 months

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 0-99 years
* Patient with neonatal intellectual disability and/or hypotonia followed at one of three inclusion centers
* Patient or parent has been informed about the study and has signed an informed consent form
* Genetic analysis by high-throughput DNA sequencing (gene panel, exome, genome) did not identify any abnormality explaining the patient's phenotype.
* If the patient's phenotype is suggestive of Prader-Willi syndrome or Angelman syndrome: a methylation anomaly test on chromosome 15 was negative.
* If the patient's phenotype is suggestive of fragile X syndrome: a repeat expansion analysis of the FMR1 gene was negative.
* If the patient's phenotype is suggestive of myotonic dystrophy type I, DM1: a repeat expansion analysis of the DMPK gene was negative.
* Patient entitled to or beneficiary of a social security scheme

Exclusion Criteria:

* Patient deprived of liberty
* Pregnant or breast-feeding woman,
* The person required to sign the consent form does not understand French
* Person under guardianship and/or curatorship

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Patients with identified deleterious variant at RNA level | Through study completion, an average of 42 month.
  The number of patients initially in diagnostic errancy in whom a deleterious variant at RNA level was identified by transcriptomic analysis (RNAseq).

SECONDARY OUTCOMES:
Comparison of the number of variants obtained from blood and from fibroblasts | Through study completion, an average of 42 month.
  Number of deleterious RNA variants identified in patients with diagnostic errancy using ARNseq on fibroblasts and deleterious RNA variants identified using ARNseq on blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance publique - hôpitaux de Marseille, Marseille, Provence-Alpes-Côt-d'Azue, France

IPD SHARING:
Plan to Share IPD: No